CLINICAL TRIAL: NCT02454023
Title: SLEep APnea Screening Using Mobile Ambulatory Recorders After TIA/Stroke (SLEAP SMART): A Randomized Controlled Trial
Brief Title: SLEep APnea Screening Using Mobile Ambulatory Recorders After TIA/Stroke
Acronym: SLEAP SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 116-2015
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Stroke; Transient Ischemic Attack; Obstructive Sleep Apnea
Keywords: Stroke; Transient ischemic attack; Obstructive sleep apnea; Portable sleep monitor; Screening
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (Active Comparator): Patients receive usual standard of care for investigating obstructive sleep apnea after stroke/transient ischemic attack, which is in-laboratory polysomnography.
  Interventions: Device: In-laboratory polysomnography
- Portable sleep monitor (ApneaLink Air) (Experimental): Patients will undergo screening for obstructive sleep apnea using the ApneaLink Air portable sleep monitor.
  Interventions: Device: Portable sleep monitor (ApneaLink Air)

INTERVENTIONS:
Device: Portable sleep monitor (ApneaLink Air) — Use of a portable sleep monitor that records respiratory effort, pulse, oxygen saturation and nasal flow, and reports apneas, hypopneas, flow limitation, snoring and blood oxygen saturation in order to detect obstructive sleep apnea.
  Arms: Portable sleep monitor (ApneaLink Air)
Device: In-laboratory polysomnography — Level 1 in-laboratory polysomnography for the detection of obstructive sleep apnea.
  Arms: Standard of care

SUMMARY:
Obstructive sleep apnea (OSA) is common after stroke/TIA and, left untreated, is associated with recurrent vascular events, poor functional outcomes, and long-term mortality. Despite its high prevalence, OSA often remains underdiagnosed after stroke. The purpose of this study is to evaluate portable sleep monitors (PSMs) as a broad screening tool for OSA after stroke/TIA. The study investigators hypothesize that the screening with PSMs will lead to an increase in the diagnosis of treatable OSA after stroke/TIA and an improvement in sleep-related and functional outcomes.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is common after stroke and, left untreated, is associated with recurrent vascular events, poor functional outcomes, and long-term mortality. Despite its high prevalence, OSA often remains underdiagnosed after stroke. While in-laboratory polysomnography studies are the gold standard for diagnosing OSA, their use is limited by the lack of availability, patient unwillingness to sleep overnight at a laboratory and high costs. Home-based PSMs can accurately diagnose OSA and are much more accessible, convenient and low-priced compared to in-laboratory sleep studies.

The primary purpose of this study is to determine whether broad screening for OSA using PSMs, as compared to usual care, increases the proportion of patients diagnosed with treatable OSA after stroke or TIA. Secondary aims include whether screening with PSMs increases the proportion of patients treated for OSA with continuous positive airway pressure (CPAP) and whether functional outcomes and sleep-related outcomes are improved. Finally, the study will also determine whether this approach is cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Imaging-confirmed stroke or stroke-neurologist diagnosed TIA in the past 6-months, and
* Outpatients being managed at the Sunnybrook Stroke Prevention clinic or inpatients on the Sunnybrook Stroke Unit.

Exclusion Criteria:

* Prior diagnosis of OSA
* Current use of CPAP
* Life expectancy less than 12 months
* The presence of conditions known to compromise the accuracy of portable sleep monitoring, such as moderate to severe pulmonary disease or congestive heart failure
* Oxygen therapy (eg. nasal prongs), a nasogastric tube, or other medical devices that would interfere with the placement of the sensors of the sleep monitoring device and/or CPAP
* Physical impairment, aphasia, or language barrier restricting ability to complete study assessments, overnight sleep monitoring, and/or comply with CPAP therapy, and no caregiver available to assist the patient with the study requirements
* Facial or bulbar weakness or trauma restricting the ability to create a seal with a CPAP mask
* Pregnancy
* Occupation that would make randomization to the standard of care arm unethical
* Not covered by Ontario health insurance plan (OHIP)
* Unable to attend follow-up assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients diagnosed with treatable OSA | 6 & 12 months
  Proportion of patients diagnosed with treatable OSA by 6 & 12 months

SECONDARY OUTCOMES:
Proportion of patients prescribed CPAP for treatable OSA | 6 & 12 months
  Proportion of patients prescribed CPAP for treatable OSA by 6 & 12 months
Cost to deliver each management strategy and treatment | 6 months
  Cost to deliver each management strategy and treatment by 6 months
Sleep-related quality of life (Functional Outcomes of Sleep Quality questionnaire) | 6 months
  Sleep-related quality of life (Functional Outcomes of Sleep Quality questionnaire) at 6 months
Daytime sleepiness (Epworth Sleepiness Scale) | 6 & 12 months
  Daytime sleepiness (Epworth Sleepiness Scale) at 6 & 12 months
Neurological outcomes (as assessed by the Stroke Impact Scale) | 6 months
  Neurological outcomes (as assessed by the Stroke Impact Scale) at 6 months
Neurological outcomes (as assessed by the modified Rankin scale) | 6 months
  Neurological outcomes (as assessed by the modified Rankin scale) at 6 months
Neurological outcomes (as assessed by the National Institutes of Health stroke scale) | 6 months
  Neurological outcomes (as assessed by the National Institutes of Health stroke scale) at 6 months
24-hr ambulatory blood pressure | 6 months
  24-hr ambulatory blood pressure at 6 months
New vascular events (stroke, TIA, myocardial infarction, coronary artery stenting) | 12 months
  Assessed via telephone call at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark I Boulos, MD, MSc, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Boulos MI, Colelli DR, Vaccarino SR, Kamra M, Murray BJ, Swartz RH. Using a modified version of the "STOP-BANG" questionnaire and nocturnal oxygen desaturation to predict obstructive sleep apnea after stroke or TIA. Sleep Med. 2019 Apr;56:177-183. doi: 10.1016/j.sleep.2018.12.021. Epub 2019 Jan 7. PMID 30803829
- [Result] Colelli DR, Kamra M, Rajendram P, Murray BJ, Boulos MI. Predictors of CPAP adherence following stroke and transient ischemic attack. Sleep Med. 2020 Feb;66:243-249. doi: 10.1016/j.sleep.2018.10.009. Epub 2018 Oct 24. PMID 30522873
- [Derived] Veitch MR, AlHamid MA, Muir RT, Dharmakulaseelan L, Ramirez JR, Gao F, Swartz RH, Murray BJ, Black SE, Boulos MI. Association between cerebral small vessel disease and periodic limb movements of sleep in patients with stroke/TIA. Sleep. 2025 Apr 11;48(4):zsaf027. doi: 10.1093/sleep/zsaf027. PMID 39901803
- [Derived] Boulos MI, Kamra M, Colelli DR, Kirolos N, Gladstone DJ, Boyle K, Sundaram A, Hopyan JJ, Swartz RH, Mamdani M, Loong D, Isaranuwatchai W, Murray BJ, Thorpe KE. SLEAP SMART (Sleep Apnea Screening Using Mobile Ambulatory Recorders After TIA/Stroke): A Randomized Controlled Trial. Stroke. 2022 Mar;53(3):710-718. doi: 10.1161/STROKEAHA.120.033753. Epub 2021 Oct 11. PMID 34628939
- [Derived] MacDonald AA, Rajendram P, Kamra M, Murray BJ, MacDonald PA, Boulos MI. Predictors of in-laboratory polysomnography attendance in a cohort of patients with stroke or TIA. Sleep Med. 2020 Feb;66:159-164. doi: 10.1016/j.sleep.2019.10.002. Epub 2019 Oct 14. PMID 31877507